CLINICAL TRIAL: NCT02557360
Title: Effectiveness of S-adenosyl-L-methionine in Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Laval University (Other)
Responsible Party: Principal Investigator, Wunsch Ewa, MD, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/02/A/NZ5/00321
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Primary Biliary Cirrhosis
Keywords: liver injury; detoxification; S-adenosyl-L-methionine; quality of life
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S-adenosyl-L-methionine (Experimental): Patients with primary biliary cirrhosis will be treated with S-adenosyl-L-methionine, tablets 800 mg twice a day (daily dosage 1600 mg) for six months
  Interventions: Dietary Supplement: S-adenosyl-L-methionine

INTERVENTIONS:
Dietary Supplement: S-adenosyl-L-methionine — Patients will be treated with S-adenosyl-L-methionine, tablets 800 mg twice a day (daily dosage 1600 mg) for six months

SUMMARY:
Primary biliary cirrhosis (PBC) is a chronic cholestatic liver disorder which may lead to several symptoms such as intractable pruritus or chronic fatigue, significantly impairing patients quality of life. Recent studies show, that chronic liver diseases are associated with an acquired deficiency of S-adenosyl-L-methionine (SAMe) synthetase, responsible for the synthesis of SAMe from methionine. SAMe deficiency is associated with impaired detoxification and hepatoprotection and exacerbate liver injury. Supplementation with SAMe has proven useful in several liver diseases.

The study group will include 20 patients with PBC diagnosed with European Association for the Study of the Liver (EASL) criteria, who have been already treated with ursodeoxycholic acid (UDCA). They will receive SAMe in the dose of 1600 mg bd over the period of 6 months. Both clinical and laboratory aspects will be analyzed: liver serum biochemistry, serum and urine bile acids metabolites, transient elastography and health related quality of life.

DETAILED DESCRIPTION:
Background: Primary biliary cirrhosis is a chronic cholestatic liver disorder which may lead to end stage liver disease causing death or requiring liver transplantation. Additionally, a significant proportion of patients suffers from complications related to impaired bile secretion such as intractable pruritus, chronic fatigue, osteoporosis or lipid disturbance. They all have a significant consequence for patients well being, quality of life and economical aspects of health care systems. Pathogenesis of PBC remains to be fully elucidated. Recent studies show,that chronic liver diseases are associated with an acquired deficiency of S-adenosyl-L-methionine synthetase, an enzyme responsible for the synthesis of SAMe from methionine. SAMe initiates two very important protective metabolic pathways: transmethylation and transsulphuration. As a result of the later, glutathione, taurine and sulphate group are synthesized. Thus SAMe deficiency is associated with impaired detoxification and hepatoprotection and exacerbate liver injury. Supplementation with SAMe has proven useful in alcoholic liver disease, obstetric cholestasis and elimination of hepatitis C virus (HCV). The investigators' studies on experimental models where cholestasis was induced in vitro with lithocholic acid and 17-beta estradiol glucuronide showed that supplementation with SAMe exerts a significant anticholestatic effect. Interestingly, simultaneous administration of SAMe and ursodeoxycholic acid (UDCA) exerts an additive effect.

Methods: The study group will include 20 patients PBC diagnosed with EASL criteria, who have been already treated with UDCA. They will receive UDCA in the dose of 13 - 15mg/kg bw plus SAMe in the dose of 1600 mg bd over the period of 6 months.

The key aim of the project is to analyze the effect of SAMe on the health related quality of life and liver biochemistry. Blood and urine samples (from 24hr urine collection) will be collected for liver biochemistry and metabolites of bile acids. Additionally transient elastography will be performed before and after 6 months SAMe treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary biliary cirrhosis diagnosed with EASL criteria;
* treatment with UDCA at least 3 months.

Exclusion Criteria:

* overlap syndromes (i.e. autoimmune hepatitis), viral hepatitis;
* decompensated liver cirrhosis (Child-Pugh class B-C);
* other diseases that can affect quality of life and mood: decompensated diabetes mellitus, renal insufficiency requiring dialyses, malignancy, heart failure ≥ New York Heart Association (NYHA) II, rheumatoid arthritis, asthma, mood disorders, depression;
* treatment with: steroids, statins, rifampicin, antidepressants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
PBC-40 questionnaire | 6 months
  Questionnaire consists 40 questions in 5 domains: Cognition, Itch, Fatigue, Social-Emotional and Other Symptoms, marked with a five-point scale (1=never to 5=always), with higher scores denoting greater symptoms impact and poorer quality of life. The possible range of each domain were: Other Symptoms domain 7-35, Itch 3-15, Fatigue 11-55, Cognitive 6-30, Social and Emotional 13-65 points.

SECONDARY OUTCOMES:
Liver fibrosis measured by transient elastography | 6 months
  To analyse the influence of SAMe treatment on liver stiffness
Number of participants with abnormal laboratory values (liver biochemistry) | 6 months
  To analyse the influence of SAMe treatment on liver function parameters
Number of participants with changes in bile acids pool | 6 months
  To analyse the influence of SAMe treatment on 17 bile acids metabolites in serum and urine

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Wunsch, Szczecin
  - Milkiewicz, Warsaw

REFERENCES:
- [Derived] Wunsch E, Raszeja-Wyszomirska J, Barbier O, Milkiewicz M, Krawczyk M, Milkiewicz P. Effect of S-adenosyl-L-methionine on liver biochemistry and quality of life in patients with primary biliary cholangitis treated with ursodeoxycholic acid. A prospective, open label pilot study. J Gastrointestin Liver Dis. 2018 Sep;27(3):273-279. doi: 10.15403/jgld.2014.1121.273.icz. PMID 30240471